CLINICAL TRIAL: NCT02044445
Title: Is the IVF Outcome Dependent on the Time Interval Between hCG Administration and Oocyte Retrieval?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Assistant Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHR-10
Record Dates: First submitted 2013-10-10; First posted 2014-01-24 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Subfertility
Keywords: IVF, hCG, oocyte retrieval, time interval
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 36 h group (Active Comparator): Oocyte retrieval will be performed 36 hours after hCG administration
  Interventions: Procedure: Oocyte retrieval will be performed 36 h or 38 h after hCG administration
- 38 h group (Active Comparator): Oocyte retrieval will be performed 38 hours after hCG administration
  Interventions: Procedure: Oocyte retrieval will be performed 36 h or 38 h after hCG administration

INTERVENTIONS:
Procedure: Oocyte retrieval will be performed 36 h or 38 h after hCG administration — Oocyte retrieval will be performed 36 h or 38 h after hCG administration
  Other Names: oocyte retrieval at 36 hours following hCG administration; oocyte retrieval at 38 hours following hCG administration

SUMMARY:
During controlled ovarian hyperstimulation (COH), human chorionic gonadotrophin (hCG) is administered to trigger the final follicular maturation before oocyte retrieval, in an attempt to mimic the physiologic effects of LH. The hCG is administered when more than three follicles ≥17mm in mean diameter have developed.

The time interval between hCG administration and oocyte retrieval is of critical importance since the time after luteinizing stimulus is a period of intense processes including the start of luteinization, expansion of cumulus cells and oocyte meiotic maturation.

The commonly practiced hCG administration time of 33 to 36 h in most IVF cycles aims to avoiding spontaneous ovulation before oocyte retrieval. However, several studies have shown that significantly more high quality embryos have been obtained with a prolonged hCG-to-oocyte interval of 38 h. It has been hypothesized that longer interval would be beneficial in improving oocyte quality and achieving optimal maturation.

Currently there are no data on the effect of the time interval between hCG administration and oocyte retrieval on IVF outcome in GnRH antagonist cycles. The aim of this study is to determine whether there is any difference in in vitro fertilization outcome when oocyte retrieval takes place at 36 h or 38 h following hCG administration

ELIGIBILITY:
Inclusion Criteria:

* women undergoing fresh IVF cycle with recombinant FSH and GnRH antagonists
* regular spontaneous menstrual cycle (24-35 days)
* age ≤ 43 years
* FSH ≤ 20 IU/L

Exclusion Criteria:

* History of previous ovarian surgery
* Women with Stage III-IV Endometriosis
* Women undergoing natural cycle IVF

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2009-11; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
retrieval rate (cumulus-oocyte complexes/ follicles> 11 mm) | up to 38 h after hCG administration

SECONDARY OUTCOMES:
Clinical pregnancy rate (evidence of intrauterine sac with fetal heart activity at 6-8 weeks of gestation) | At 6-8 weeks of gestation
Total number of oocytes retrieved | up to 38 h after hCG administration

CONTACTS AND LOCATIONS:
Locations (1):
- Unit for Human Reproduction, 1st Dept of Obstetrics and Gynaecology, Medical School, Aristotle University of Thessaloniki, Thessaloniki, Greece